CLINICAL TRIAL: NCT06252220
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind First in Human, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DA-1726 in Participants With Obesity.
Brief Title: First in Human Study in Subjects With Obesity, But Otherwise Healthy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DA-1726-1001
Record Dates: First submitted 2024-01-09; First posted 2024-02-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking is to be done at the pharmacy level. The pharmacists that do not have other responsibilities in the study will prepare and administer the drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 - Single Ascending Dose (Active Comparator): Single doses of DA-1726 in adult participants (aged 18 to 65 years) with obesity (BMI ≥30 - 45 kg/m2). DA-1726 will be administered via subcutaneous (SC) injection within the clinic setting.
  Interventions: Drug: DA-1726; Drug: Placebo to DA-1726
- Part 2 - Multiple Ascending Dose (Placebo Comparator): Multiple doses of DA-1726 in adult participants (aged 18 to 65 years) with obesity (BMI ≥30 - 45 kg/m2). DA-1726 will be administered via subcutaneous (SC) injection within the clinic setting.
  Interventions: Drug: DA-1726; Drug: Placebo to DA-1726

INTERVENTIONS:
Drug: DA-1726 — Active
Drug: Placebo to DA-1726 — Placebo

SUMMARY:
This is a First in Human study to evaluate the safety and tolerability of DA-1726 following single and multiple doses in participants with obesity, but otherwise healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, placebo-controlled, double-blind, sequential parallel group study to investigate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple ascending doses of DA-1726 in adult participants (aged 18 to 65 years) with obesity (BMI ≥30 - 45 kg/m2). DA-1726 will be administered via subcutaneous (SC) injection within the clinic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent prior to initiation of any study specific procedures/activities.
2. Males and females ≥18 to <=65 years of age, at the time of signing informed consent, who have been diagnosed with obesity, or have signs/symptoms consistent with obesity.
3. Except for obesity, otherwise healthy as determined by the investigator based on a medical evaluation including physical exam, medical history, laboratory tests, and ECGs.
4. Body mass index (BMI) ≥ 30 kg/m2 to 45 kg/m2 (Obesity to be confirmed by Caliper test).
5. Has maintained a stable body weight during the 3 months prior to Screening (<5% body weight change).
6. Willing to maintain current diet and physical activity regimen.

   * SAD Cohorts (Be willing to eat a standard diet while in the Clinical Research Unit).
   * MAD Cohorts (Be willing to eat a standard diet while in the Clinical Research Unit). If appetite decreases, participants may not maintain their current diet.
7. Females must be of non-reproductive potential:

   * Postmenopausal defined as:

     * Age of ≥55 years with no menses for at least 12 months; OR
     * Age <55 years with no menses for at least 12 months AND with a follicle-stimulating hormone level >40 IU/L or according to the definition of "postmenopausal range" for the laboratory involved; OR
   * History of hysterectomy; OR
   * History of bilateral oophorectomy
   * History of tubal ligation (surgically sterile)
8. Males must agree to practice an acceptable method of effective birth control while on study through 5 half-lives plus one week after receiving last dose of DA-1726.

Acceptable methods of birth control include:

* Sexual abstinence
* Vasectomy and testing that shows there are no sperm in semen.
* Condom with spermicide (male) in combination with barrier methods (diaphragm, cervical cap, or cervical sponge), hormonal birth control, or IUS (females)

Exclusion Criteria:

1. History or clinical evidence of diabetes mellitus, including a fasting glucose of ≥ 120 mg/dL and/or HbA1c ≥ 6.5% at Screening.
2. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2).
3. History of cholecystectomy < 6 months prior to screening.
4. Subjects with screening calcitonin level of ≥15 pg/mL (calcitonin levels will be monitored during the study).
5. Triglycerides ≥500 mg/dL at Screening.
6. History of pancreatitis.
7. Have a medical history or current evidence of clinically significant cardiac condition as evidenced by any of the following at Screening :

   * QTc at Screening from locally generated data of >450 msec in males or >470 msec in females or history of long QT syndrome
   * Supine systolic BP higher than 150 mmHg and a supine diastolic BP higher than 95 mmHg at Screening or check-in
   * Supine HR of <50 or >100 beats per minute on 2 of 3 triplicate ECGs at Screening or check-in
   * Heart block of the 1st, 2nd, or 3rd degree
   * Sick sinus syndrome (irregular heartbeat patterns)
   * Disorders in cardiac conduction
   * Peripheral blood circulation issues
   * Heart valve conditions
   * Cardiomyopathy
   * History of myocardial infarction
   * Unstable angina
   * History of heart artery bypass surgery
   * History of stroke
   * History of heart failure
8. Regular consumption of caffeine-containing beverages, including coffee, tea, energy drinks, and caffeinated sodas, exceeding 3 cups per day.
9. Current use of tobacco products or having a history of tobacco use within the past 6 months.
10. Have significant previous or current history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data.
11. History of GI abnormality that could affect GI motility (including small bowel or colonic resection, inflammatory bowel disease, irritable bowel syndrome, gastroparesis [clinically significant gastric emptying abnormality], and colon / GI tract cancer).
12. Have a history of chronic medical conditions involving the heart, liver, or kidneys (e.g., atherosclerotic coronary vascular disease (ASCVD), heart failure, liver cirrhosis, chronic kidney disease).
13. Untreated or uncontrolled hypo/hyperthyroidism defined as thyroid-stimulating hormone >6 mIU/L or <0.4 mIU/L.
14. Obesity that was induced by other endocrinologic disorders (e.g., Cushing's Syndrome).
15. Evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies.
16. Evidence of hepatitis C and/or positive hepatitis C antibody and hepatitis B, hepatitis B core antibody, and/or positive hepatitis B surface antigen.
17. Have a history or presence of psychiatric disorders that would present a safety risk or may significantly impair the participant's ability to comply with study procedures.
18. Any lifetime history of a suicidal attempt or any suicidal behavior, as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS).
19. History of malignancy of any type, other than basal cell carcinoma, occurring less than 5 years prior to randomization.
20. History of substance abuse (i.e., alcohol or illicit substances) within 12 months prior to Screening; and/or a positive test for alcohol/drugs of abuse at Screening.
21. Previous surgical treatment for obesity or any form of bariatric surgery.
22. Currently receiving treatment in another investigational drug or device study or 5 half lives or 30 days since last dose of investigational drug, whichever is longer.
23. Participants with a history of significant allergic or drug reactions (NSAIDs or antibiotics) or known allergy to DA 1726 excipients that would place them at increased risk.
24. Have received any vaccine ≤30 days prior to check-in.
25. Albumin level <3.5 g/dL (<35 g/L) at Screening.
26. Aspartate aminotransferase (AST) ≥1.25 × upper limit of normal (ULN) at Screening.
27. Alanine aminotransferase (ALT) ≥1.25 × upper limit of normal (ULN) at Screening.
28. Bilirubin >1.25 upper limit of normal (ULN) at Screening.
29. Absolute neutrophil count <lower limit of normal (LLN) at Screening.
30. Estimated glomerular filtration rate of ≤60 mL/min for women and men (based on the Chronic Kidney Disease Epidemiology Collaboration equation) at the Screening.
31. Fasting low-density lipoprotein ≥160 mg/dL at Screening.
32. Hemoglobin <LLN at Screening.
33. Platelet count <LLN at Screening.
34. Current or history of treatment with medications that may cause significant weight gain, within 3 months of Screening, including:

    * Systemic corticosteroids (except for a short course of treatment, i.e., 7-10 days)
    * Tricyclic antidepressants
    * Atypical antipsychotics
    * Mood stabilizers (e.g., imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid and its derivatives, and lithium)
    * Antidiabetic Medications (e.g., insulin or certain sulfonylureas, that may lead to weight gain)
    * Beta-blockers (e.g., the ones used to treat conditions like hypertension that may cause weight gain)
    * Antihistamines (particularly the first-generation ones, that may have sedative effects and could potentially contribute to weight gain)
    * Contraceptives
    * Any non-steroidal anti-inflammatory drugs
35. Current participation (or within the last 3 months) in an organized weight reduction program or currently using or has used within 3 months prior to Screening: pramlintide, sibutramine, orlistat, zonisamide, topiramate, phentermine, naltrexone, lorcaserin, liraglutide, semaglutide, tirzepatide or metformin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From date of randomization (baseline) until the discontinuation or completion, whichever came first, assessed up to 26 Days for Part 1 and 47 Days for Part 2.
  AEs, SAEs, TEAEs and AEs leading to treatment discontinuation.

SECONDARY OUTCOMES:
Pharmacokinetic | From date of randomization (baseline) until the discontinuation or completion, whichever came first, assessed up to 26 Days for Part 1 and 47 Days for Part 2.
  PK profile of DA-1726 serum concentrations of DA-1726 over time.
Immunogenicity | From date of randomization (baseline) until the discontinuation or completion, whichever came first, assessed up to 26 Days for Part 1 and 47 Days for Part 2.
  Measurement of anti-drug antibodies and neutralizing antibodies at baseline and at identified points during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No